CLINICAL TRIAL: NCT02203708
Title: Effect on Relationship of a Brief Preventive Program: Pragmatic Pilot Randomized Controlled Trial." - Supportive Program for Mother With BPD
Brief Title: Supportive Program for Mother With BPD
Acronym: PAM-B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 11 199 08; Interregional PHRC 2011 (Other Grant/Funding Number: French Ministry of Health)
Record Dates: First submitted 2013-01-22; First posted 2014-07-30 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2014-07

CONDITIONS: Parent-child Problem; Borderline Personality Disorder
Keywords: BPD (Borderline Personality Disorder); Mother/child
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BPD prevention (Active Comparator): Supportive Program for Mother with BPD (SuPMother-B) : BPD mothers participate to prevention program in groups or/and house calls.
  Interventions: Other: Supportive Program for Mother with BPD (SuPMother-B).
- Usual care of BPD mothers (No Intervention): BPD mothers don't participate to Supportive Program (SuPMother-B).

INTERVENTIONS:
Other: Supportive Program for Mother with BPD (SuPMother-B). — The development of the program is based on several principles: group process, groupware, mentalization, parental values, behavioral strategies and information on the child's needs, knowledge of the BPD and the strategies of get better. The program will last 10 sessions of group of about 2h.
  Minimal intervention. All study participants receive an individual interview about 45 minutes with a psychiatrist for three objectives: information on the diagnosis of BPD, information on resources for health care and educational aids.
  Arms: BPD prevention

SUMMARY:
Borderline Personality Disorder (BPD) is characterized by a pervasive pattern of instability of interpersonal relationships, self-image and emotions as well as marked impulsivity. When patients have children, they are at high risk of severe emotional and relational disturbances (withdrawal, low self-esteem, depression, suicidal thoughts). In addition, studies support the effectiveness of parental guidance group to reduce emotional and behavioral difficulties of children. To our knowledge there are no programs directed to mothers with BPD who received a controlled evaluation.

From experience with parental guidance, data from the observation of children of patients with BPD and psychosocial programs directed to patients BPD, we have built for preventive intervention. The Supportive Program for Mothers with BPD (SuPMother-B) consists of 10 group sessions providing information (education, childcare, care specific to BPD) and promotes mother-child interactions (observation, games).

Purpose: Compare the effect of a program (SuPMother-B) group, of 10 sessions, offered to mothers with a BPD in addition to a minimal intervention (diagnostic announcement and provision of health care resources) on behavior withdrawal of children at 6 months compared to a group of mothers receiving only minimal intervention.

Primary outcome: Difference at 6 months between the experimental and control groups on scores on the assessment scale withdrawal (Alarm Distress Baby (ADBB)).

ELIGIBILITY:
Inclusion Criteria:

Mother:

* Women with children and at least one child aged 2 months to 2 years, Borderline Personality Disorder with SIDP (Structured Interview for DSM Personality Disorders)
* age above 18 years
* written consent

Child:

* ages between 2 months and 2 years,
* parental consent for research participation.

Exclusion Criteria:

Mother:

* chronic psychotic disorder, major depressive disorder, current mania or hypomania,
* legal protection,
* if no child can be included, the mother cannot be included.

Child :

•major psychomotor development disorder or psychiatric disorder according to the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-07; Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Difference between the experimental and control groups on scores on the assessment scale withdrawal (Alarm Distress Baby (ADBB)). | Visit 3 at 6 months

SECONDARY OUTCOMES:
Brunet-Lezine Scale | Visit 2 (inclusion), 3 (6 months) and 4 (1 year)
  This scale permits to assess the psychomotor development of the child.
Borderline Personality Disorder Severity Index (BPDSI) | Visit 2 (inclusion), 3 (6 months) and 4 (1 year)
  Borderline Personality Disorder Severity Index (BPDSI) is a semi-structured interview assessing the frequency and severity of manifestations of borderline personality disorders of the mother during an agreed period (3 months to 1 year).
Global Assessment Scale | Visit 2 (inclusion), Visit 3 (6 months), Visit 4 (1 Year)
  This scale corresponds to the 5th axis of the Diagnostic and Statistical Manual of Mental Disorders (DSM) and permits to assess the overall functioning of the mother.
Difference between the experimental and control groups on scores on the assessment scale withdrawal (Alarm Distress Baby (ADBB)). | Visit 2 (inclusion) and visit 4 (1 Year)
M.I.N.I. 5.0.0 French version | Visit 2 (inclusion), Visit 3 (6 months), Visit 4 (1 year)
  Structured interview to assess 17 disorders such as actual or passed depression, mania, abuse...
Parenting Sense of Competence Scale (P.S.O.C) | Visit 2 (inclusion), Visit 3 (6 months), Visit 4 (1 year)
  This scale assess the perceived competence of the parent's role as educator.
social and demographic data | Visit 2 (inclusion), Visit 3 (6 months), Visit 4 (1 year)
  marital status, profession, socio-economic level, number of children
Data on care pathways | Visit 2 (inclusion), Visit 3 (6 months), Visit 4 (1 year)
  Questionnaire established by the research team to evaluate the use of care services by the mothers and children.

CONTACTS AND LOCATIONS:
Overall Officials: CHEYNIER, Principal Investigator — UTAMS PMI Empalot; LATOUR, Principal Investigator — UTAMS PMI Reynerie; BLEY-RIBET, Principal Investigator — UTAMS PMI Bonnefoy; MULQUIN, Principal Investigator — UTAMS PMI Rangueil; KOUBAA, Principal Investigator — UTAMS PMI Cazères; BERTIN, Principal Investigator — UTAMS PMI Montauban
Locations (1):
- Service de psychiatrie de l'enfant et de l'adolescent - Hôpital La Grave - centre Hospitalier de Toulouse, Toulouse, France